CLINICAL TRIAL: NCT06801132
Title: The Effectiveness of an Online Self-Delivered Death Anxiety Intervention: a Pilot Randomized Controlled Trial
Brief Title: The Effectiveness of an Online Self-Delivered Death Anxiety Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: 101 Institute, Ministry of Civil Affairs of the People's Republic of China (Unknown)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Facing death anxiety pilot
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Death Anxiety
Keywords: Death Anxiety; randomized controlled trial; self-delivered
MeSH Terms: conditions — Necrophobia | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization was conducted by an independent research assistant, and the random sequence was concealed from the investigator until the process was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Death anxiety (Experimental)
  Interventions: Behavioral: Online self-delivered death anxiety intervention
- Waiting-List (WL) condition (Other): Participants assigned to WL will be asked not to use our death anxiety intervention or seek additional help related to death anxiety during the 1-week intervention period. After the one-month follow-up of the experimental group, the WL group will receive the same intervention for death anxiety. WL participants will also be given contact information to use in case of increasing distress.
  Interventions: Behavioral: Waiting-List (WL) condition

INTERVENTIONS:
Behavioral: Online self-delivered death anxiety intervention — The online self-guided death anxiety intervention developed in this study is based on the Death Education and CBT framework. It took approximately two hours to complete the full intervention. The main content includes:
  1. Emotional reactions and behavioral manifestations about death, fear management theories, and Chinese cultural attitudes toward death;
  2. Imagine what you would like to say to yourself at the end of your life, and learn about various attitudes towards death through numerous examples;
  3. Expressive writing, with moderate emotional exposure to stimulate reflection, accompanied by breathing exercises and positive thinking about death, to improve tolerance and control of death anxiety, and finally to correct biased perceptions by examining bad beliefs about death;
  4. Prioritize the importance of things and make a practical action plan to enrich your life.
  Arms: Death anxiety
Behavioral: Waiting-List (WL) condition — Participants assigned to WL will be asked not to use our death anxiety intervention or seek additional help related to death anxiety during the 1-week intervention period. After the one-month follow-up of the experimental group, the WL group will receive the same intervention for death anxiety. WL participants will also be given contact information to use in case of increasing distress.
  Arms: Waiting-List (WL) condition

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of the online self-delivered death anxiety intervention developed by our team in the general population with a randomized controlled trial. The study will recruit 50 participants, with 25 randomized to the death anxiety intervention group and 25 randomized to the control group (waiting list). The online intervention on death anxiety consists of 4 phases that take about 2 hours in total. The primary outcome DAS (Death Anxiety Scale) and DABBS (Death Anxiety Beliefs and Behaviors Scale) will be administered on baseline, post-treatment, 1-month follow-up, and 3-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Normal literacy skills and ability to use a smartphone proficiently
* Higher death anxiety that is above the cutoff of our measurement
* Voluntarily participate in this intervention and be able to provide informed consent.

Exclusion Criteria:

* Severe depressive state or risk of suicidal self-injury, i.e., the total score of Patient Health Questionnaire 9-item ≥19 or the score of 9th item ≥2
* Diagnosed within 6 months with schizophrenia, depression, bipolar disorder, and other psychiatric disorders
* Have received any intervention for death anxiety or CBT intervention on any topic within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Templer Death Anxiety Scale (T-DAS) | baseline, post treatment(1 week), 5 weeks, 13 weeks
  The T-DAS consists of 15 items, describing the experiences that individuals feel when facing death. The Chinese version suggests a 5-point scale according to the later extended version of the scale, ranging from 1 "Strongly Agree" to 5 "Strongly Disagree", with higher scores representing more severe death anxiety. The higher the score, the more serious the death anxiety, and a total score greater than 43 according to the rules can be considered to have a high level of death anxiety. The Chinese version of T-DAS has been widely used and has shown good reliability and validity.
Death Anxiety Beliefs and Behaviors Scale (DABBS) | baseline, post treatment(1 week), 5 weeks, 13 weeks
  The DABBS consists of 18 entries describing overall feelings about death (4 entries), thoughts and beliefs related to death (7 entries), and avoidance behaviors related to death (7 entries), with the scale being scored on a 5-point scale ranging from 1, "Strongly Disagree/Never Have This Thought/Never Avoid This Behavior" to 5 "Strongly agree/always have this thought/always avoid this behavior," with higher scores representing the severity of the individual's adverse beliefs and behaviors regarding death.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9-item | baseline, post treatment(1 week), 5 weeks, 13 weeks
  Patient Health Questionnaire 9-item (PHQ-9), a self-report measure for depressive symptoms in the past two weeks, comprises 9 items rated from 0 (not at all) to 3 (nearly every day). The PHQ-9 has good psychometric properties in Chinese adolescents.
Generalized Anxiety Disorder 7-item | baseline, post treatment(1 week), 5 weeks, 13 weeks
  Generalized Anxiety Disorder 7-item (GAD-7) scale is a 7-item self-report measure to assess anxiety symptoms in the past two weeks. Each item is rated from 0 (not at all) to 3 (nearly every day). The Chinese version GAD-7 score has good psychometric properties among adolescents.
Insomnia Severity Index (ISI) | baseline, post treatment(1 week), 5 weeks, 13 weeks
  The ISI consists of seven items that assess the severity of subjective insomnia in the past two weeks, including, for example, difficulty in falling asleep, sleep satisfaction, impairment of daytime functioning, etc. The total score ranges from 0-28, with higher scores representing more severe insomnia. The Chinese version of ISI has been shown to have good reliability and validity.
4-dimensional anxiety scale | baseline, post treatment(1 week), 5 weeks, 13 weeks
  This is a 40-item scale for measuring multi-dimensional anxiety, which includes 4 dimensions (emotional, physiological, cognitive, and behavioral) and 9 subscales (emotional, psychosomatic, autonomic, general cognitive, phobia, over-committed, repetitive, social, and avoidance). The higher the score on this scale, the more severe the anxiety in a certain area.
Ryff's Psychological Well-being Scale (PWS) | baseline, post treatment(1 week), 5 weeks, 13 weeks
  The short version used in this study contains 18 entries, including six dimensions of positive relations, autonomy, environmental mastery, personal growth, purpose in life, and self-acceptance. The six dimensions of self-acceptance are scored on a 6-point scale ranging from 1 "not at all" to 6 "very much", with higher scores representing higher psychological well-being. The Chinese version of PWS has been translated by Taiwanese scholars and has been proven to have Good reliability and validity.

OTHER OUTCOMES:
Adverse Childhood Experiences | baseline
  An adverse childhood experiences questionnaire measuring the adverse childhood experiences with 13 items. A higher number of adverse childhood experiences represents worse childhood experiences.
Social support | baseline, 5 weeks
  The 12-item Multidimensional Scale of Perceived Social Support (score from 1 to 7, and total score varies from 12 to 84). A higher score represents better social support.
Post-traumatic responses scale - Flight subscale | baseline, post treatment(1 week), 5 weeks, 13 weeks
  This is a 9-item subscale measuring flight responses of the Post-traumatic responses scale, which is a 5-point Likert scale (score from 0 to 4, and total score varies from 0 to 36). A higher score represents a higher post-traumatic avoidance tendency.
Irritability | baseline, post treatment(1 week), 5 weeks, 13 weeks
  A 17-item irritability measurement scale, the Peking irritability scale, measures impulsive emotions, thoughts, and behaviors on a 5-point Likert scale (score from 1 to 5, and total score varies from 17 to 85). A higher score represents higher irritability.
A sense of stability | baseline, post treatment(1 week), 5 weeks, 13 weeks
  A 7-item 6-point Likert scale that measures the subjective feeling of being settled and fulfilled in one's current life. The higher the score on the scale, the stronger the sense of stability.
Alexithymia | baseline, post treatment(1 week), 5 weeks, 13 weeks
  A 23-item Peking alexithymia scale measures thoughts and behaviors that prevent people from feeling or recognizing negative emotions on a 5-point Likert scale (1 to 5, and total scores vary from 23 to 115). A higher score represents more severe alexithymia.
Emotion regulation | baseline, post treatment(1 week), 5 weeks, 13 weeks
  An 18-item cognitive emotion regulation questionnaire measures the ability of emotion regulation on a 5-point Likert scale (1 to 5, and total scores vary from 18 to 90). A higher score represents better emotion regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No